CLINICAL TRIAL: NCT07225582
Title: Development of Optimal Sensory Feedback Strategies to Maximize Function After Tetraplegia: A Sub-study of the Reconnecting the Hand and Arm to the Brain (ReHAB) Clinical Trial
Brief Title: Development of Optimal Sensory Feedback Strategies to Maximize Function After Tetraplegia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other); Cleveland Clinic Lerner Research Institute (Unknown)
Responsible Party: Principal Investigator, Emily Graczyk, Assistant Professor, Biomedical Engineering, Case Western Reserve University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY20190226; R01HD117313 (NIH)
Record Dates: First submitted 2025-11-04; First posted 2025-11-06 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injury Cervical; Spinal Cord Injuries (Complete and Incomplete)
Keywords: spinal cord injury; tetraplegia; intracortical microstimulation; peripheral nerve stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia | interventions — Brain-Computer Interfaces; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Intracortical microstimulation and peripheral nerve stimulation for people with tetraplegia (Experimental): The purpose of the proposed study is to investigate the perception and functional impact of sensory neurostimulation in participants with tetraplegia. Investigators will develop and implement novel paradigms of intracortical microstimulation (ICMS) applied to primary somatosensory cortex (S1) and peripheral nerve stimulation (PNS) applied to upper extremity nerves through chronically-implanted cuff electrodes. Investigators will also develop and assess hybrid neurostimulation paradigms involving paired application of ICMS and PNS. For each paradigm, investigators will quantify the perceived sensation with classic psychophysical methods. Investigators will also implement the approach into closed-loop tasks in virtual reality controlled through decoded cortical signals recorded from intracortical microelectrode arrays. Finally, investigators will assess the impact of each stimulation paradigm on residual sensory function.
  Interventions: Device: Brain Computer Interface (BCI) - Functional Electrical Stimulation (FES) system

INTERVENTIONS:
Device: Brain Computer Interface (BCI) - Functional Electrical Stimulation (FES) system — Participants with tetraplegia who have received intracortical arrays in the sensory cortex and peripheral nerve cuff electrodes will undergo a variety of stimulation paradigms to investigate the perception and functional impact of sensory neurostimulation.

SUMMARY:
The goal of this clinical trial is to learn more about how stimulating the nerves involved in sensation (either in the limbs or in the brain) can be used to restore sensation in participants who have a spinal cord injury. Participants in this study will have already been enrolled in the "Reconnecting the Hand and Arm to the Brain (ReHAB)" study, and received small electrodes in a part of the brain that is involved in sensing touch and pressure in the hand. The ReHAB study participants will also have received electrodes around the nerves in their arm. In this clinical trial, participants will receive two types of electrical stimulation:

* Intracortical microstimulation (ICMS) which involves sending small electrical pulses to the part of the brain that processes sensation.
* Peripheral nerve stimulation (PNS) which involves sending small electrical pulses to the nerves in the arm that transmit sensations from the hand.

Researchers will try different patterns of stimulation for both ICMS and PNS and study how the participants perceive the sensations from the different stimulation patterns. The researchers will also study how combining ICMS and PNS affects the perceived sensations.

DETAILED DESCRIPTION:
The overall goal of this study is to compare the sensations that are perceived from intracortical microstimulation (ICMS) to those perceived from peripheral nerve stimulation (PNS), and also to perceived sensations from a combination of ICMS and PNS.

Preceding study

Participants for this study will be individuals with a high-level spinal cord injury who are already enrolled in the "Reconnecting the Hand and Arm to the Brain (ReHAB)" clinical trial (ID# NCT03898804). The ReHAB clinical trial involves receiving tiny electrode arrays in the brain and small electrodes around some of the nerves in the arm. The goal of the ReHAB clinical trial is to restore arm and hand movement and sensation in individuals with paralysis from a spinal cord injury.

Goals of this clinical trial

The purpose of the proposed study is to investigate the perception and functional impact of sensory neurostimulation in participants with tetraplegia. Investigators will develop and implement novel paradigms of ICMS applied to primary somatosensory cortex (S1) and PNS applied to upper extremity nerves through chronically-implanted cuff electrodes. Investigators will also develop and assess hybrid neurostimulation paradigms involving paired application of ICMS and PNS. For each paradigm, investigators will quantify the perceived sensation with classic psychophysical methods. Investigators will also implement the approach into closed-loop tasks in virtual reality controlled through decoded cortical signals recorded from intracortical microelectrode arrays. Finally, investigators will assess the impact of each stimulation paradigm on residual sensory function.

In Aim 1, investigators will develop a novel ICMS paradigm that attempts to reproduce both the temporal and spatial activation patterns that occur in S1 during normal touch. Investigators will compare this novel paradigm to other existing ICMS encoders. Investigators will assess the impact of each ICMS encoder on perceptual response, task performance in virtual reality (VR), and residual sensory function. In Aim 2, investigators will develop novel PNS paradigms and assess the efficacy of PNS for sensory feedback in people with tetraplegia for the first time. As in Aim 1, investigators will develop and compare several PNS encoders, including those that reproduce aspects of the peripheral response to normal touch and traditional linear encoders. We will assess the impact of each PNS encoder on perceptual response, task performance in VR, and residual sensory function. In Aim 3, we will develop hybrid neurostimulation paradigms that pair ICMS with PNS. We will assess the impact of stimulation encoder and stimulation amplitude on the perceived sensations generated by hybrid stimulation. We will then investigate the impact of PNS-ICMS timing delays within the hybrid neurostimulation paradigm on the perceptual response, functional impact, and impact on residual sensory function.

All participants will participate in all aims and will receive all stimulation approaches and perform all tasks and measures. All participants will serve as their own control for the planned statistical analyses. The study will generate tens of thousands of perceptual response data points, hundreds of functional task data points, and hundreds of thousands of intracortical recordings (for exploratory analyses).

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in the ReHAB clinical trial and received ReHAB system components via implantation surgery.
2. Willingness and availability to follow the study protocol.

Exclusion Criteria:

1. Lack of function or operability of all implanted ReHAB system components
2. Severe pain or other chronic medical condition that would prevent the participant from completing study-related activities

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Force matching success rate | From enrollment to around two years after enrollment
  Percentage of force matching trials per block in which the target force was achieved before the time limit
Object discrimination accuracy | From enrollment to around two years after enrollment
  Percentage of trials per block in which the correct object was identified
Discrimination threshold | From enrollment until around two years post-enrollment
  Minimal change in stimulation that results in a reliably distinguishable change in perceived magnitude
Tactor detection threshold | From enrollment to around two years after enrollment
  Minimal mechanical stimulus, delivered by a tactor that the participant can reliably perceive

SECONDARY OUTCOMES:
Sensory dynamic range | From enrollment until around two years post-enrollment
  Difference in minimum and maximum stimulation levels that elicit detectable, comfortable sensation
Projected field location | From enrollment until around two years post-enrollment
  The position of the sensory percept reported on a hand/arm diagram
Sensation quality | From enrollment to around two years after enrollment
  The participant's description of the quality of the sensation evoked by stimulation, reported as a selection of descriptor words
Naturalness rating | From enrollment until around two years post-enrollment
  The participant's rating of the perceived naturalness of the stimulus on an open-ended scale
Tactor discrimination threshold | From enrollment to around two years after enrollment
  Minimal change in mechanical touch input that results in a reliably distinguishable change in perceived magnitude
Force matching time to target | From enrollment to around two years after enrollment
  The time elapsed from the go cue required for the participant to hit the force target
Posture matching success rate | From enrollment to around two years after enrollment
  Percentage of posture matching trials per block in which the target posture was achieved before the time limit

CONTACTS AND LOCATIONS:
Overall Officials: Emily Graczyk, Ph.D., Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD may be shared for publications.

REFERENCES:
- See also: This website provides information about the ReHAB Study. — https://rehabstudy.org